CLINICAL TRIAL: NCT00152321
Title: Strategies Targeting Osteoporosis to Prevent Recurrent Fractures (STOP# Study)
Brief Title: Strategies Targeting Osteoporosis to Prevent Recurrent Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sumit R. Majumdar, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Alberta; CIHR-MOP #62906
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Osteoporosis; Fractures
Keywords: osteoporosis; wrist fractures; quality improvement; knowledge translation
MeSH Terms: conditions — Osteoporosis; Fractures, Bone; Wrist Fractures | interventions — Educational Status; Counseling; Physicians

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Multifaceted intervention
  Interventions: Behavioral: Patients (education, counseling) and Physicians (reminders,1-page guidelines).; Behavioral: Multifaceted intervention
- B (Active Comparator): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Patients (education, counseling) and Physicians (reminders,1-page guidelines).
  Arms: A
Behavioral: Multifaceted intervention — Educational materials, counseling, opinion leader based guidelines, reminders
  Arms: A
Other: Usual Care
  Arms: B

SUMMARY:
An evidence-based quality improvement intervention will overcome multiple barriers to best practice and improve rates of diagnosis and effective treatment for osteoporosis in high-risk patients. The intervention will be directed at patients (education and counseling) and their primary care physicians (reminders and opinion leader generated and endorsed single page guidelines)

DETAILED DESCRIPTION:
Background: Osteoporosis leads to decreased bone mass, skeletal fragility, and fractures. Fractures cause disability, deformity, and even death. Osteoporosis affects 1.4 million Canadians, 25% of women and 12% of men >50 years. Current guidelines recommend aggressive secondary prevention in patients with osteoporosis and a fracture, because risk of re-fracture is as high as 20% within a year, and because treatment can reduce this risk by 40-50%. Because bisphosphonates are safe and efficacious in preventing both vertebral and nonvertebral fractures, they are the treatment of choice. Patients with a wrist fracture are ideally suited to a strategy of case-finding and secondary prevention since this is a sentinel event in the natural history of osteoporosis: wrist fractures are common and easily diagnosed, always present to medical attention, are usually related to low bone mass, and wrist fractures tend to occur years before the more devastating fractures of the hip or vertebrae. However, these patients are under-diagnosed and under-treated. Eight studies have reported that one year after a wrist fracture, fewer than 10-20% of patients >50years of age have been tested or treated for osteoporosis. A significant care gap between evidence-based best practice and usual care exists.

Objective: To improve the quality of care for patients with osteoporosis and wrist fractures.

Hypothesis: An evidence-based quality improvement intervention will overcome multiple barriers to best practice and improve rates of diagnosis and effective treatment for osteoporosis in high-risk patients. The intervention will be directed at patients (education and counseling) and their primary care physicians (reminders and opinion leader generated and endorsed single page guidelines).

Specific Aims: To determine whether the proposed intervention can:

Aim #1- Increase use of effective osteoporosis treatment in patients with a fracture of the wrist.

Aim #2- Increase rates of bone mineral density testing in these patients.

Aim #3- Increase osteoporosis-related knowledge in these patients.

Aim #4- Increase satisfaction with medical care in these patients.

Study Design: A prospective randomized controlled trial comparing the proposed intervention to usual care in Emergency Departments and Fracture Clinics. Eligible patients will be >50 years and present with any wrist fracture and not be taking bisphosphonates. Primary outcome is the proportion of patients starting bisphosphonate treatment within 6 months of fracture. The main secondary outcomes are starting any effective osteoporosis treatment (bisphosphonates, calcitonin, raloxifene, or hormone replacement therapy) and bone mineral density testing within 6 months. There will be blinded ascertainment of all outcomes. The intervention is expected to increase the primary outcome (bisphosphonate treatment) by at least 20% over usual care rates of 10%. With an alpha=0.05, beta=0.90, and a 20% loss to followup, the minimum required sample size is 220 patients.

ELIGIBILITY:
Inclusion Criteria:

All patients 50 years of age or older with a wrist fracture who present to the Emergency Departments or Fracture Clinics at our two study sites will be eligible for study enrollment. Specifically:

1. Age 50 years or greater,
2. Any distal forearm fracture

Exclusion Criteria:

1. Unable to give simple informed consent,
2. Unwilling to participate in the study,
3. Unable to understand, read, or converse in English,
4. Place of residence outside Capital Health or longterm care facility,
5. Already receiving osteoporosis treatment with a bisphosphonate,
6. Previously documented allergy or intolerance to a bisphosphonate,
7. Currently enrolled in the pilot study or other osteoporosis study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2003-09; Primary Completion 2006-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients starting bisphosphonate treatment within 6 months of fracture | 6 months

SECONDARY OUTCOMES:
Appropriate care (BMD test performed and treatment if low bone mass) | 6 months
Bone mineral density testing | 6 months
Self reported diagnosis of osteoporosis and other knowledge | 6 months
Satisfaction with care | 6 months
Health related quality of life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sumit R Majumdar, MD, MPH, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Majumdar SR, Johnson JA, McAlister FA, Bellerose D, Russell AS, Hanley DA, Morrish DW, Maksymowych WP, Rowe BH. Multifaceted intervention to improve diagnosis and treatment of osteoporosis in patients with recent wrist fracture: a randomized controlled trial. CMAJ. 2008 Feb 26;178(5):569-75. doi: 10.1503/cmaj.070981. PMID 18299546
- [Result] Majumdar SR, Lier DA, Rowe BH, Russell AS, McAlister FA, Maksymowych WP, Hanley DA, Morrish DW, Johnson JA. Cost-effectiveness of a multifaceted intervention to improve quality of osteoporosis care after wrist fracture. Osteoporos Int. 2011 Jun;22(6):1799-808. doi: 10.1007/s00198-010-1412-1. Epub 2010 Sep 29. PMID 20878389
- [Derived] Majumdar SR, Johnson JA, Bellerose D, McAlister FA, Russell AS, Hanley DA, Garg S, Lier DA, Maksymowych WP, Morrish DW, Rowe BH. Nurse case-manager vs multifaceted intervention to improve quality of osteoporosis care after wrist fracture: randomized controlled pilot study. Osteoporos Int. 2011 Jan;22(1):223-30. doi: 10.1007/s00198-010-1212-7. Epub 2010 Apr 1. PMID 20358359